CLINICAL TRIAL: NCT05109832
Title: A Clinical Trial of the Absorption, Metabolism, and Excretion of [14C]IMP4297 in Chinese Adult Male Healthy Volunteers - A Human Material Balance and Biotransformation Study of [14C]IMP4297
Brief Title: A Study of Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]IMP4297 to China Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMP4297-109
Record Dates: First submitted 2021-10-12; First posted 2021-11-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 14C-IMP4297 (Experimental): In this study, one 100 mg dose of 14C IMP4297 Oral Suspension, 100 mg (100 μCi).
  Interventions: Drug: 14C-IMP4297

INTERVENTIONS:
Drug: 14C-IMP4297 — 14C marked IMP4297

SUMMARY:
A Phase I, Open-label Study of Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]IMP4297 Following a Single Oral Dose to China Healthy Male Subjects

DETAILED DESCRIPTION:
Study design A Phase I, single-center, open-label, single arm study is designed to evaluate Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]IMP4297 Following a Single Oral Dose to China Healthy Male Subjects.

6-8 subjects are planned to be enrolled (at least 6 subjects complete the study)

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet all of the following inclusion criteria to be included in the study:

  1. Volunteers must fully understand the objective, nature, methods and possible adverse reactions of the trial, volunteer to be volunteers, and sign an informed consent form before the start of any study procedures, and at the same time guarantee that the volunteers will personally participate in the study during any procedures.
  2. Chinese healthy male volunteers aged between 18 and 55 (including cut-off values) at the time of screening.
  3. Volunteers with a body mass index (BMI) of 18.0-28.0 kg/m2 (including cut-off values), and a body weight of ≥ 50.0 kg.

Exclusion Criteria:

* Volunteers who meet any of the following criteria cannot be included in this study:

  1. Diseases with abnormal clinical manifestations that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bones.
  2. A history of allergic diseases (including drug allergies and food allergies, etc.).
  3. A history of any gastrointestinal diseases that will affect drug absorption such as dysphagia, irritable bowel syndrome, and inflammatory bowel disease; active hemorrhoids or perianal diseases accompanied by regular/current blood in the stool; habitual constipation or diarrhea.
  4. Those who have undergone surgery within 3 months before screening, or who plan to undergo surgery during the study period, and those who have undergone surgery that will affect drug absorption, metabolism, or excretion.
  5. Those who cannot tolerate venipuncture, and those who have a history of needke sickness and blood phobia.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum concentration) | 3 months
  peak concentration
Tmax | 3 months
  Time to peak
AUC0-inf (Area under the curve from time 0 to infinity) | 3 months
  area under the curve from time zero to infinity
AUC0-last (Area under the curve from time 0 to the last time with quantifiable concentration) | 3 months
  AUC0-last area under the curve from time zero to the time with the last quantifiable concentration
t½ (Elimination half-life) | 3 months
  elimination half-life
CL/F (Apparent clearance) | 3 months
  apparent clearance
Vz/F (apparent volume of distribution ) | 3 months
  apparent volume of distribution
urine and fecal samples for quantification analysis | 3 months
  Assessment of recovery percent in urine and feces by liquid chromatography-radiochemical-detection。 Get Percent (%) of each radiolabeled drug-related material will be determined in urine and feces
After oral administration of [14C] IMP4297 in healthy volunteers, radioactive metabolite spectrogram are obtained to identify the main metabolites and clarify the main biotransformation pathways. | 3 months
  Proportion of different metabolites，Assessment of metabolites (metabolites identification and main metabolites) in plasma/urine/faeces by liquid chromatography-radiochemical-detection

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No